CLINICAL TRIAL: NCT04530383
Title: A Randomized, Double-blind, Crossover Clinical Trial of Metformin in Those With CFRD on CFTR Modulator Therapy to Improve Ion Channel Function
Brief Title: Effects of Metformin on Airway Ion Channel Dysfunction in Cystic Fibrosis-related Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Matthias Salathe, MD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00146063
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis-related Diabetes; Cystic Fibrosis
Keywords: Metformin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin dose regimen A (Experimental): Participants with CFRD on elexacaftor/tezacaftor/ivacaftor who meet criteria and agree to participation in the study will be placed on metformin 500 mg twice daily on study week 0 after undergoing study procedures through week 14. They will then undergo a two week washout period. For the second half of the study metformin will be resumed and, if tolerated, dose will be increased by 500mg on weeks 17 and 18 to a final dose of 1000 mg twice daily through end of study (week 30).
  Interventions: Drug: Metformin Hydrochloride
- Metformin dose regimen B (Experimental): Participants with CFRD on elexacaftor/tezacaftor/ivafactor who meet criteria and agree to participation in the study will be placed on metformin 500 mg twice daily on study week 0 after undergoing study procedures. If tolerated, dose will be increased by 500mg on weeks 1 and 2 to a final dose of 1000 mg twice daily through week 14.They will then undergo a two week washout period. For the second half of the study metformin will be resumed at a dose of 500 mg twice daily through the end of study (week 30).
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — 500-1000 mg twice daily
  Other Names: Glucophage

SUMMARY:
The purpose of this study is to assess the efficacy of metformin to improve airway ion channel function in those with CF-related diabetes (CFRD)

DETAILED DESCRIPTION:
Up to 30 patients with CFRD on highly effective CFTR modulator therapy who meet criteria and agree to participation in the study will be placed on metformin 500mg twice daily (low) and 1000mg twice daily (normal) in a randomized order (simple randomization). There will be a dose-escalation with each dosing regimen starting with 500mg twice daily for a week, followed by 500mg in the AM and 1000mg in the PM for another week and finally followed by 1000mg twice daily until the end of normal dose cycle (in those in the normal dose portion of the crossover trial). A matching placebo pill will be utilized so participants do not know which dosing regimen, low or normal, they are on during each 14-week period. Participants will continue each dosing regimen of metformin for 14 weeks with a washout period of 2 weeks between dose changes. To minimize risk of B12 deficiency, a known side effect of long-term metformin use, we will also provide a supplement of 1000 µg oral cyanocobalamin daily for the duration of the trial.

ELIGIBILITY:
Inclusion criteria:

1. Age >18 years with a prior diagnosis of CF.
2. Use of ivacaftor or elexacaftor/tezacaftor/ivacaftor for 30 days prior to day 0
3. 3. Diagnosis of CFRD with evidence of continued glucose intolerance at least 6 months after starting elexacaftor/tezacaftor/ivacaftor will be based upon one of the following:

   1. Insulin use
   2. Hemoglobin A1C >6.5%
   3. Fasting glucose >126 mg/dl
   4. Non-fasting glucose >200 mg/dl (random or as part of a 2-hr OGTT)

Exclusion criteria:

1. Prior lung or liver transplant
2. Use of supplemental oxygen
3. BMI <18
4. CF pulmonary exacerbation requiring hospitalization or intravenous antibiotics in the preceding 30 days
5. Systemic corticosteroid or regular non-steroidal anti-inflammatory use in the preceding 30 days
6. Cardiac, renal (creatinine clearance <45 mL/minute), neurologic, psychiatric, endocrine or neoplastic diseases that are judged to interfere with participation in the study
7. Alanine aminotransferase, aspartate aminotransferase or alkaline phosphatase >1.5X the upper limit of normal; bilirubin >3 mg/dL
8. Taking medications that interact with metformin.
9. Vitamin B12 deficiency
10. Pregnancy or lactation
11. Inability or unwillingness to comply with an approved contraceptive method during the study period (females of childbearing age)
12. Use of medications known to be strong CYP inducers or moderate to strong CYP inhibitors
13. In the opinion of the investigator any severe or acute or chronic condition or laboratory abnormality that may increase the risk associated with trial participation or make the subject inappropriate for enrollment
14. Participation in another interventional trial that, in the opinion of the investigator, has the potential to affect the primary outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change in BK channel gene expression | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Levels of LRRC26 (big potassium channel regulatory subunit) mRNA will be measured by polymerase chain reaction from nasal cells acquired via brushing

SECONDARY OUTCOMES:
Change in BK function, as measured by nasal potential difference testing | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Nasal potential difference testing measures direct BK current in the nasal epithelium, with greater current indicating greater BK function
Change in receptor for receptor for advanced glycation end products (RAGE) gene expression | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Levels of RAGE mRNA will be measured by polymerase chain reaction from nasal cells acquired via brushing
Change in advanced glycation end products (AGE) | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Plasma levels of AGE, receptor for AGE (RAGE), soluble RAGE and S100A12 will be quantified by ELISA
Change in sweat chloride | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Measured as a secondary marker of CFTR function, with lower levels indicating greater CFTR function
Change in lung function | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Measured by percent predicted forced expiatory volume in one second captured on spirometry (FEV1)
Change in Quality of Life (CFQ-R) | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Measured by Patient Reported Outcome measurement tool called CFQ-R (validated)
Change in airway inflammatory markers | Baseline through week 14 and week 16 through week 30 of metformin treatment
  Inflammatory markers (interleukin-1beta, interleukin-6, interleukin-8, transforming growth factor beta1, tissue necrosis factor-alpha, matrix metalloproteinase-9 and cyclooxygenase-2) collected from nasal fluid will be measured by enzyme linked immunosorbent assay (ELISA)
Safety of metformin | Baseline through week 30 of metformin treatment
  Number of adverse events during study period
Pharmacokinetics of metformin | Week 14 and week 30 of metformin treatment
  Plasma levels of metformin will be quantified by liquid chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Salathe, M.D., Principal Investigator — Professor
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No